CLINICAL TRIAL: NCT06046807
Title: Determine the Proportion of Patients With Disabling Post Thrombotic Syndrome (Moderate or Severe) in the Long Term Within the Cohort of Patients Who Participated in the Trial CELEST Therapy.
Brief Title: Long-Term Post Thrombotic Syndrome Assessment (CELEST Long Term).
Acronym: CELEST-LT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laboratoires Innothera (Industry)
Collaborators: Floralis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A00528-37
Record Dates: First submitted 2023-09-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Post Thrombotic Syndrome
Keywords: Post thrombotic syndrome; Elastic compression stockings; long-term follow-up; Deep vein Thrombosis
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 35mmHg ECS: Subjects with first proximal DVT allocated to wear 35 mmHg elastic compression stockings (ECS) for 2 years during the CELEST RCT
  Interventions: Other: Phone call
- 25mmHg ECS: Subjects with first proximal DVT allocated to wear 25 mmHg elastic compression stockings (ECS) for 2 years during the CELEST RCT
  Interventions: Other: Phone call

INTERVENTIONS:
Other: Phone call — This follow-up will be conducted over the phone and by mail (some questionnaire may be sent by patient, as per his/her preference)

SUMMARY:
The CELEST Long term is a prospective study, assessing the very long term risk of post thrombotic syndrome (PTS) in patients enrolled in the CELEST double-blind RCT. All patients enrolled in CELEST RCT will benefit from a 7-year follow-up visit conducted over the phone. The primary objective is to assess the proportion of patients with moderate-severe PTS assessed with the patient reported Villalta score and the 2 main secondary objectives are to assess predictors of moderate to severe PTS and the impact of initial compression stockings strength (25mmHg vs. 35mmHg) on the development of moderate-severe PTS. Up to 288 patients may participate.

The investigators believe that this study has the potential to significantly improve the knowledge on the epidemiology of burdensome PTS and on the impact of different initial compression stockings strengths on the risk of PTS.

DETAILED DESCRIPTION:
The CELEST double blind RCT demonstrated that 25mmHg elastic compression stockings (ECS) were non inferior to 35mmHg ECS to prevent post thrombotic syndrome (PTS) 2 years after a first proximal deep vein thrombosis (DVT). Likely because of lack of statistical power the investigators were not able to demonstrate that 25mmHg ECS were superior in the overall RCT population and that 35mmHg ECS were superior in patients optimally adherent to ECS. Furthermore, few data are available on the very long term (>5 years).

The CELEST Long term is a prospective study, assessing the very long term risk of PTS in patients enrolled in the CELEST RCT. All patients enrolled in CELEST RCT and willing to participate are eligible and will benefit from a 7-year follow-up visit conducted over the phone.

Primary objective is to assess the proportion of patients with moderate-severe PTS defined as a patient reported Villalta score (PRVS) ≥10 or a venous leg ulcer ipsilateral to index DVT. Secondary objectives include predictors of moderate to severe PTS, impact of initial ECS strength on the development of moderate-severe PTS, impact of anticoagulant treatment (type and duration) on the development of moderate to severe PTS, proportion of PTS (defined as PRVS≥5 or ipsilateral leg ulcer) and impact of PTS on patient's QOL. Study should last 1 year and up to 288 patients may participate.

The investigators believe that this study has the potential to significantly improve the knowledge on the epidemiology of burdensome PTS and on the impact of different initial CE strengths on the risk of PTS.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled and followed in the CELEST RCT*

Exclusion Criteria:

* Patients who withdrew consent or died during the 2-year follow-up of the CELEST RCT.
* Patients who decline or are unable to participate (including severe memory loss issues) to the long-term follow-up

  * CELEST RCT main inclusion/exclusion criteria were: adult (>18 years at time of enrolment) patients first unilateral acute symptomatic proximal lower limb DVT

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were enrolled in the CELEST RCT
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2023-12-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with moderate-severe PTS in the whole cohort | At the phone follow-up up to 3 months
  PTS defined with the patient reported Villalta score (PRVS). Moderate-severe PTS: PRVS≥10 or presence of a venous leg ulcer in the leg ipsilateral to index DVT
  The Villalta score consists in 11 questions (5 on subjective symptoms and 6 on objective signs).
  Each question is coded between 0 and 3 (0: none - 1: mild - 2: moderate - 3: severe). The total score is the sum of the 11 questions and therefore ranges from 0 to 33, where a high value indicates a high level of disability.
  An additional question asks about the presence of ulcers. If the calculated score is < 15, a value of 15 is assigned to the ulcer score.
  The thresholds used are as follows:
  * presence of PTS if Villalta ≥ 5
  * presence of disabling PTS (moderate, severe) if Villalta ≥ 10
  * presence of severe PTS if Villalta ≥ 15

SECONDARY OUTCOMES:
Predictors of moderate-severe PTS | Since enrolment in the CELEST CRT
  Predictors of moderate-severe PTS in the whole cohort
Impact of initial ECS strength on the development of moderate-severe PTS | Since enrollment in the CELEST study
  Comparison of proportion of moderate-severe PTS between patients randomized in the 25mmHg ECS vs. 35mmHg ECS group
Impact of initial type of ECS on the development of moderate-severe PTS | Since enrollment in the CELEST study
  Comparison of proportion of moderate-severe PTS between patients who chose to wear above knee vs. below knee ECS during CELEST RCT
Impact of adherence to RCT's ECS on the development of moderate-severe PTS | Since enrollment in the CELEST study
  Comparison of proportion of moderate-severe PTS according to adherence to ECS during CELEST RCT
Assessment of the use of ECS after the end of the RCT in terms of use, strength, length, adherence, duration | Since enrolment in the CELEST study with focus on the period end of RCT to long-term follow-up
  Description of the use of ECS among study participants since the end of their participation in the CELEST RCT
Factors influencing the the decision to continue, stop or resume ECS | During the 2-year celest study and during the long-term follow-up
  Description of the reasons that led to the decision to continue, stop or resume ECS
Impact of anticoagulant treatment on the development of moderate-severe PTS | During the 2-year celest study and during the long-term follow-up
  Comparison of proportion of moderate-severe PTS according to type and duration of anticoagulant treatment during CELEST RCT
Proportion of patients with any PTS | At the phone follow-up up to 3 months
  PTS present if PRVS≥5 or presence of a venous leg ulcer in the leg ipsilateral to index DVT
Predictors of any PTS | At the phone follow-up up to 3 months
  Predictors of PTS (defined as a PRVS≥5 or presence of a venous leg ulcer in the leg ipsilateral to index DVT) in the whole cohort
Proportion of patients who developed a serious adverse events (SAE) in the cohort | During the 2-year celest study and during the long-term follow-up
  SAEs assessed are death, venous thromboembolic recurrence, major bleeding and peripheral arterial disease. SAEs are defined according to the International Society on Thrombosis and Haemostasis criteria. These events will be adjudicated by the study adjudication committee
Impact of PTS on patients' quality of life | At the phone follow-up up to 3 months
  Comparison of QOL scores according to the presence or absence of PTS and its severity; QOL will be assessed using CIVIQ-20 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc Bosson, MD, PhD, Principal Investigator — University Grenoble Alpes, France; Jean Philippe Galanaud, MD, PhD, Principal Investigator — University of Toronto, Canada
Locations (1):
- ROLLAND, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided
Relevant deidentified participant data (with a data dictionary) will be available to other researchers on reasonable request after publication, approval from both principal investigators and sponsor, and after a data access agreement is signed

REFERENCES:
- [Background] Ten Cate-Hoek AJ. Lower strength stockings: is less better? Lancet Haematol. 2022 Dec;9(12):e865-e866. doi: 10.1016/S2352-3026(22)00266-6. No abstract available. PMID 36455603
- [Background] Utne KK, Ghanima W, Foyn S, Kahn S, Sandset PM, Wik HS. Development and validation of a tool for patient reporting of symptoms and signs of the post-thrombotic syndrome. Thromb Haemost. 2016 Jan;115(2):361-367. doi: 10.1160/th15-04-0318. Epub 2015 Sep 17. PMID 26422814
- [Background] Ageno W, Squizzato A, Wells PS, Buller HR, Johnson G. The diagnosis of symptomatic recurrent pulmonary embolism and deep vein thrombosis: guidance from the SSC of the ISTH. J Thromb Haemost. 2013 Aug;11(8):1597-602. doi: 10.1111/jth.12301. No abstract available. PMID 23682905
- [Background] Kaatz S, Ahmad D, Spyropoulos AC, Schulman S; Subcommittee on Control of Anticoagulation. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Nov;13(11):2119-26. doi: 10.1111/jth.13140. No abstract available. PMID 26764429
- [Background] Kraaijpoel N, Tritschler T, Guillo E, Girard P, Le Gal G. Definitions, adjudication, and reporting of pulmonary embolism-related death in clinical studies: A systematic review. J Thromb Haemost. 2019 Oct;17(10):1590-1607. doi: 10.1111/jth.14570. Epub 2019 Jul 31. PMID 31301689
- [Background] Launois R, Reboul-Marty J, Henry B. Construction and validation of a quality of life questionnaire in chronic lower limb venous insufficiency (CIVIQ). Qual Life Res. 1996 Dec;5(6):539-54. doi: 10.1007/BF00439228. PMID 8993100
- [Background] Makedonov I, Kahn SR, Galanaud JP. Prevention and Management of the Post-Thrombotic Syndrome. J Clin Med. 2020 Mar 27;9(4):923. doi: 10.3390/jcm9040923. PMID 32230912
- [Background] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Result] Galanaud JP, Genty-Vermorel C, Barrellier MT, Becker F, Jabbour V, Blaise S, Bura-Riviere A, Comte A, Grange C, Guenneguez H, Maufus M, Ouvry P, Richaud C, Rolland C, Schmidt J, Sevestre MA, Verriere F, Bosson JL; CELEST trial investigators. 25 mm Hg versus 35 mm Hg elastic compression stockings to prevent post-thrombotic syndrome after deep vein thrombosis (CELEST): a randomised, double-blind, non-inferiority trial. Lancet Haematol. 2022 Dec;9(12):e886-e896. doi: 10.1016/S2352-3026(22)00247-2. PMID 36455606
- [Result] Galanaud JP, Genty-Vermorel C, Rolland C, Comte A, Ouvry P, Bertaina I, Verriere F, Bosson JL. Compression stockings to prevent postthrombotic syndrome: Literature overview and presentation of the CELEST trial. Res Pract Thromb Haemost. 2020 Oct 30;4(8):1239-1250. doi: 10.1002/rth2.12445. eCollection 2020 Nov. PMID 33313464